CLINICAL TRIAL: NCT01428245
Title: Assessment of Sensitivity of the Hypothalamic GnRH Pulse Generator to Estradiol and Progesterone Inhibition in Early Pubertal Girls (JCM026)
Brief Title: Assessment of Sensitivity of the Hypothalamic GnRH Pulse Generator to Estradiol and Progesterone Inhibition
Acronym: JCM026
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The research questions was changed/de-prioritized. Only one subject completed.
Sponsor: University of Virginia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, John Marshall, Director, Center for Research in Reproduction, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14100; U54HD028934 (NIH); P50HD028934 (NIH)
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Results first posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Hyperandrogenemia; Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Progesterone; Estradiol; Estrogens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Progesterone, estrace (Experimental): oral progesterone suspension (20 mg/ml, 25-100 mg) three times a day at 0700, 1500, and 2300 hr to achieve mean plasma concentrations over the range of 2-8 ng/ml for seven days
  oral estrace, 0.5-1 mg once a day for seven days
  Interventions: Drug: Progesterone; Drug: Estrace (estrogen)

INTERVENTIONS:
Drug: Progesterone — oral progesterone suspension (20 mg/ml, 25-100 mg) three times a day at 0700, 1500, and 2300 hr for seven days
Drug: Estrace (estrogen) — oral estrace, 0.5-1 mg once a day for seven days
  Other Names: estradiol

SUMMARY:
Gonadotropin-releasing hormone (GnRH) is a hormone that regulates the ability of the pituitary to secrete two hormones, luteinizing hormone (LH) and follicle-stimulating hormone (FSH). LH and FSH control the production of female hormones (such as estrogen and progesterone) and the development of eggs by the ovary. Progesterone and estrogen then decrease the number of GnRH pulses produced by the brain (and therefore the number of LH pulses from the pituitary). The ability to decrease GnRH pulses seems to be very important for normal menstrual function in adult women. The purpose of this study is to learn more about how GnRH and LH pulses are controlled during puberty. The information gathered in this study will hopefully allow us to learn more about how menstrual cycles are normally established in girls during puberty.

DETAILED DESCRIPTION:
In this study, the investigators will aim to discover the effect of 7 days of estrogen and progesterone on GnRH pulses in girls in early and mid puberty. Ultimately, if the investigators understand these normal processes, the investigators may be able to better understand abnormalities of puberty.

ELIGIBILITY:
Inclusion Criteria:

* Girls ages 8 to 14
* Tanner 1-3 pubertal stage
* Pre-menarchal
* Normal screening labs

Exclusion Criteria:

* Abnormal screening labs
* Congenital adrenal hyperplasia
* Hyperandrogenism (e.g., hirsutism, elevated free testosterone level)
* Hemoglobin <12 mg/dL or hematocrit < 36% (Subjects will be offered the opportunity to take iron supplementation for 60 days if their hematocrit is slightly low (33-36%) (suggestive of iron deficiency anemia) and will then return for retesting of their hemoglobin/hematocrit.)
* Weight < 31 kg
* History of peanut allergy, deep venous thrombosis, breast cancer, endometrial cancer, or cervical cancer
* On hormonal medications (including oral contraceptive pills) or on medications known to affect the reproductive axis within 3 months of the study
* Pregnant or breast feeding
* Participation in a research study within the past 30 days that involved taking a study drug.
* Participation in a research study that involved taking up to or greater than 473 ml's of blood within the past 60 days.
* Cigarette smoking
* History of surgery that required bedrest within the past 30 days
* Family history of hypercoagulability or unexplained thromboembolic disease (not in setting of bedrest, surgery, or malignancy)
* In order to ensure an adequate number of younger girls, no more than 4 enrolled subjects will be Tanner stage 3

Ages: 8 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2011-04-22 (Actual); Primary Completion 2013-05-14 (Actual); Study Completion 2013-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C. Marshall, MD, PhD, Principal Investigator — University of Virginia
Locations (1):
- Center for Research in Reproduction, University of Virginia, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 subjects enrolled in this study. 2 subjects completed screening procedures only (these 2 subjects were withdrawn from study prior to being assigned to an arm of intervention).
Groups:
- Progesterone, Estrace: oral progesterone suspension (20 mg/ml, 25-100 mg) three times a day at 0700, 1500, and 2300 hr to achieve mean plasma concentrations over the range of 2-8 ng/ml for seven days
  oral estrace, 0.5-1 mg once a day for seven days
  Progesterone: oral progesterone suspension (20 mg/ml, 25-100 mg) three times a day at 0700, 1500, and 2300 hr for seven days
  Estrace (estrogen): oral estrace, 0.5-1 mg once a day for seven days
Period: Overall Study
Arm/Group | Progesterone, Estrace
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Progesterone, Estrace
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: LH Pulse Frequency as a Function of Day 7 Progesterone
Description: number of LH pulses per 11 hours on Day 7 of progesterone
Time Frame: 7 days following oral estrace and progesterone administration
Population: Only one subject completed study.
Measure: Number; unit: number of LH pulses/11hr
Arm/Group | Progesterone, Estrace
Number analyzed (Participants) | 1
number of LH pulses/11hr | 0

ADVERSE EVENTS:
Time Frame: 30 days post study drug intervention
Arm/Group | Progesterone, Estrace
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-02-29): https://cdn.clinicaltrials.gov/large-docs/45/NCT01428245/Prot_SAP_000.pdf
  • Informed Consent Form (2011-07-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT01428245/ICF_001.pdf